CLINICAL TRIAL: NCT02984176
Title: Simethicone and Gynecological Laparoscopies: Does it Improve Operative Field and Postoperative Pain?
Brief Title: Simethicone: Does it Improve Operative Field and Postoperative Pain?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, Kamal Mohamed Zahran, Assistant professor of Obstetrics & Gynecology, Faculty of Medicine, Consultant and vice director, Women's Health Hospital, Assiut University, Egypt, Woman's Health University Hospital, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Simethicone and laparoscopy
Record Dates: First submitted 2016-06-28; First posted 2016-12-06 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Simethicone
Keywords: Simethicone; Laparoscopies; Pain
MeSH Terms: conditions — Pain | interventions — Simethicone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simethicone (Active Comparator): Arm 1 or Group I or Simethicone 40mg. 3 tablets (one tablet after each meal) and to fast overnight the day before the operation.
  Interventions: Drug: Simethicone Tab 40 mg
- placebo (Placebo Comparator): Arm 2 or group 2 or placebo group. 3 tablets (one tablet after each meal) and to fast overnight the day before the operation.
  Interventions: Drug: Placebo Tablets

INTERVENTIONS:
Drug: Simethicone Tab 40 mg — 3 tablets of Simethicone Tab 40 mg (one tablet after each meal) and to fast overnight the day before the operation.
  Other Names: Disflatyl
  Arms: Simethicone
Drug: Placebo Tablets — 3 tablets of Placebo Tablets (one tablet after each meal) and to fast overnight the day before the operation.
  Other Names: Placebo
  Arms: placebo

SUMMARY:
Simethicone is an oral anti-foaming agent that reduces bloating, abdominal discomfort, and abdominal pain by promoting the clearance of excessive gas along the gastrointestinal tract.

The investigators objective is to evaluate the efficacy and safety of preoperative oral simethicone for bowel preparation in gynecological laparoscopies.

DETAILED DESCRIPTION:
Introduction: Simethicone is an oral antifoaming agent that reduces bloating, abdominal discomfort, and abdominal pain by promoting the clearance of excessive gas along the gastrointestinal tract.

Objective: to evaluate the efficacy and safety of preoperative oral simethicone for bowel preparation in gynecological laparoscopies.

Methods: 100 infertile women will be scheduled for laparoscopy, patients randomized to receive either Simethicone (Group I) or placebo tablets (Group II). The primary outcome measure will be the overall exposure of the surgical field and pain scoring. Assessment of the overall exposure of the surgical field was done using a five-point scale (poor, sufficient, medium, good, and excellent). Visual analog score (VAS) will be used for assessment of postoperative pain and verbal analog scoring was used for assessment of patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Infertile patients
* aged 20 - 40 years old
* scheduled for laparoscopy

Exclusion Criteria:

* Women were excluded from the study if patients had one or more of the following:

  * scar of previous operation, uterine mass, severe endometriosis, suspicion of malignancy, history of allergic reaction to study drugs, psychiatric disorders and patient refusal

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2014-08; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
five-point scale | 1 hour

SECONDARY OUTCOMES:
The degree of bowel preparation | 1 hour
VAS | 24 hours
Patient satisfaction | 24 hours

IPD SHARING:
Plan to Share IPD: Yes